CLINICAL TRIAL: NCT06821321
Title: The Effects of Plyometric or Resistance Training on Muscle and Tendon Stiffness, and Functional Performance in Older Adults
Brief Title: Power or Plyometric Training in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20241358
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Activity, Motor
MeSH Terms: conditions — Motor Activity | interventions — Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training (Other): Participants in this group will receive plyometric training for up to 12 weeks.
  Interventions: Behavioral: Plyometric Training
- Power Resistance Training (Other): Participants in this group will receive power resistance training for up to 12 weeks.
  Interventions: Behavioral: Power Training

INTERVENTIONS:
Behavioral: Plyometric Training — Participants will receive a total of twenty-four 45-minutes in-person resistance-training sessions, twice per week, using three sets of eight repetitions per set on five upper body exercises. During resistance-training participants will be allowed 1-minute rests between sets. Participants will also perform two jump training exercises on a horizontal Pilates reformer, the leg plyometric and ankle plantar plyometric jumps.
  Arms: Plyometric Training
Behavioral: Power Training — Participants will receive a total of twenty-four 45-minutes in-person training sessions, twice per week using three sets of eight repetitions per set. During training participants will be allowed 1-minute rests between sets. Exercises will include five upper-body exercises and two lower-body exercises.
  Arms: Power Resistance Training

SUMMARY:
This study will compare the effects of high-speed power resistance training or plyometric jump training on muscle stiffness, jump performance and measures of daily activity in older adults living independently in the community.

ELIGIBILITY:
Inclusion Criteria:

* Independently living
* Between 55-90 years of age

Exclusion Criteria:

* Uncontrolled cardiovascular disease that prevents participation in a training program.
* Documented HIV infection or another immunodeficiency syndrome.
* Current neuromuscular diseases that prevent exercise.
* Current musculoskeletal injury that prevents exercise.
* Incarcerated individuals
* Montreal Cognitive Assessment (MoCA) Score below 18

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Quadriceps Muscle Stiffness measured by Kilopascals | Baseline, 10 weeks
  For muscle stiffness, three images will be taken in the longitudinal view in shear wave mode to assess stiffness of the vastus lateralis, vastus medialis and rectus femoris muscles. Color-coded images with a scale from blue (soft) to red (hard) will then be generated depending on muscle stiffness. Imaging software will then convert the wave speed data into a stiffness measures called kilopascals.
Change in Triceps Surae Muscle Stiffness measured by Kilopascals | Baseline, 10 weeks
  For muscle stiffness, three images will be taken in the longitudinal view in shear wave mode to assess stiffness of the gastrocnemius lateralis, gastrocnemius medialis and soleus muscles. Color-coded images with a scale from blue (soft) to red (hard) will then be generated depending on muscle stiffness. Imaging software will then convert the wave speed data into a stiffness measures called kilopascals.
Change in Quadriceps Tendon Stiffness measured by Kilopascals | Baseline, 12 weeks
  For tendon stiffness, three images will be taken in the longitudinal view in shear wave mode to assess stiffness of the quadriceps tendon. Color-coded images with a scale from blue (soft) to red (hard) will then be generated depending on tendon stiffness. Imaging software will then convert the wave speed data into a stiffness measures called kilopascals.
Change in Patellar Tendon Stiffness measured by Kilopascals | Baseline, 12 weeks
  For tendon stiffness, three images will be taken in the longitudinal view in shear wave mode to assess stiffness of the patellar tendon. Color-coded images with a scale from blue (soft) to red (hard) will then be generated depending on tendon stiffness. Imaging software will then convert the wave speed data into a stiffness measures called kilopascals.
Change in Achilles Tendon Stiffness measured by Kilopascals | Baseline, 12 weeks
  For tendon stiffness, three images will be taken in the longitudinal view in shear wave mode to assess stiffness of the Achilles tendon. Color-coded images with a scale from blue (soft) to red (hard) will then be generated depending on tendon stiffness. Imaging software will then convert the wave speed data into a stiffness measures called kilopascals.
Changes in Stored Elastic Energy measured by joules | Baseline, 12 weeks
  For assessment of stored elastic energy, subjects will perform a Squat Jump and a Countermovement Jump on the force platform. The Squat Jump will be performed with the subject starting in a squatted position at the knee angle of approximately 90 degrees. The subject will hold that position for 1-2 s, and then jump into the air with maximal effort. For the Countermovement Jump, the subject will start in an upright position, rapidly squat down and then jump into the air with maximal effort. For both jumps, subject's hand will be held at the waist to eliminate the effect resulting from arm swing during jump performance. For each jump, three trials will be conducted with 1 min rests between trials. For safety, an experienced assistant will stand alongside each subject while performing the test to prevent injury. Energy will be measured in Joules.
Change in Gait Economy | Baseline, 12 weeks
  Gait Economy will be measured using oxygen consumption on a treadmill at each subject's usual walking speed, one-half of the maximal walking speed, and 75% of the maximal walking speed. Each bout will last 5 minutes, with a 3-minute standing rest between bouts. Oxygen consumptions for the last 2 minutes of each bout will be used to compute energy cost and determine gait economy. Gait economy will be assessed as the oxygen used at each of the three walking speeds measured in milliliters of oxygen per kilogram of body weight per minute.

SECONDARY OUTCOMES:
Change in Muscle Thickness measured in centimeters | Baseline, 12 weeks
  Three images will be taken in the longitudinal view in B-mode. Muscle thickness will be measured by drawing a perpendicular line from the deep to superficial aponeurosis at the thickest region of each muscle. The unit of measurement is centimeters.
Change in Muscle Quality measured using grayscale | Baseline, 12 weeks
  Muscle quality will be measured using a gray scale. The black and white pixels correspond to arbitrary values of 0 (darker) to 255 (lighter), with darker colors indicating more muscle and lighter colors indicating more fat.
Change in neuromuscular performance as measured by 1-repetition maximum (1RM). | Baseline, 12 weeks
  Maximal load that can be lifted in one repetition (1RM) will be assessed in both leg press and chest press exercises. The loads on the testing equipment will be increased across 5 to 7 testing repetitions. The persons 1RM will be the highest load the person can move through the range of motion of the exercise. There are no minimum or maximum scores for this test. The higher the 1RM the stronger the person is. The unit of measurement is kilograms.
Change in the Speed of the Ten-Meter Walk Test. | Baseline, 12 weeks
  The ten-meter walk test will be used to assess gait velocity. The participants will be asked to walk at usual walking speed and as quickly as possible in a straight line on a 10-m course marked at 0, 2, 8 and 10 m. On verbal command, participants will start on the 0-m mark and stop when the 10-m mark is crossed. The total time to ambulate from the 2-m mark to the 8-m mark (6 m total) will be timed to the hundredth of a second. Two trials will be performed at each speed, and the average will be documented in meters per second. One-minute recoveries will be provided between trials.
Change in Time for the Five Times Sit-to-Stand Test. | Baseline, 12 weeks
  The five-time sit-to-stand test will be used to assess functional lower body strength. The participant will sit with arms folded across the chest and the back against the chair. On a verbal command, the participant will stand up and sit down five times as quickly as possible. Timing begins at the word go and ends when the buttocks touch the chair after the fifth repetition. One practice and two testing trials will be performed. Time will be measured in seconds.
Change in Distance of the Seated Medicine Ball Throw. | Baseline, 12 weeks
  For the Seated Medicine Ball Throw, subjects will sit in an armless chair with the back against the chair back, while holding the 6-pound medicine ball against the chest.
  Subjects will then throw the ball at a perceived 45° angle as far as possible. Subjects must complete at least three practice trials; however, subjects will be allowed more trials until comfortable with the testing procedure. Upon starting the official trial, subjects will complete three separate attempts at each varying medicine ball, to nine trials in total.
  Each of the three trials within a given medicine ball test will be separated by a 1-minute rest. Distance will be measured in centimeters.
Changes in the Six-Minute Walk Test. | Baseline, 12 weeks
  The object of the test is to walk as far as possible for six minutes. The subject will walk at a normal pace around a marked course for six minutes. The subject may stop to rest and begin again at will. The distance covered indicates aerobic fitness. The further a person walks, the better the cardiovascular condition. The units are meters.
Change in the time required to complete the timed Up-and-Go Test. | Baseline, 12 weeks
  Upon verbal cue, the subject stands up, walks around a cone placed three meters from the front edge of the chair and then returns to a seated position as quickly as possible. Time is measured in seconds.
Change in neuromuscular performance as measured by Watts | Baseline, 12 weeks
  This test measures the power a person can produce at maximal speed using loads of 20%, 40%, 60%, 80%, and 90% of 1RM for the chest press and leg press. Power shows how fast a person can do work. Unit of measure is Watts.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No